CLINICAL TRIAL: NCT05750654
Title: Effectiveness of Small Phlebotomy Tubes in Reducing Blood Transfusions in Adult Medical Intensive Care Unit and Intermediate Care Unit Patients With Anemia: A Randomized Controlled Trial
Brief Title: Effectiveness of Small Phlebotomy Tubes in Reducing Blood Transfusions in Adult Medical Intensive Care Unit and Intermediate Care Unit Patients With Anemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Javier Barreda Garcia, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSC-MS-22-1045
Record Dates: First submitted 2023-02-10; First posted 2023-03-02 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Anemia
Keywords: Blood transfusion
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Small Tube Group (Experimental)
  Interventions: Device: Small Phlebotomy Tube Group
- Standard Tube Group (Active Comparator)
  Interventions: Device: Standard Phlebotomy Tube Group

INTERVENTIONS:
Device: Small Phlebotomy Tube Group — In the small tubes group, the recommended blood volumes are 0.5 mL for hematology and single chemistry tests, and 1 mL when multiple chemistry tests are needed. A, a "non-formulary medication" order will be placed in the electronic medical record to alert nurses to collect blood in small tubes. Participants will continue to use small tubes anytime they are in the ICU or IMU.
  Arms: Small Tube Group
Device: Standard Phlebotomy Tube Group — In the standard tubes group, the recommended blood volumes are 4.0 mL for hematology and 3.0 for chemistry tests.
  Arms: Standard Tube Group

SUMMARY:
The purpose of this study is to evaluate the effectiveness of small phlebotomy tubes to reduce RBC transfusions in medical intensive care unit (ICU) and Intermediate care unit (IMU) patients with low hemoglobin compared with standard size tubes, to compare the intervention and the control groups in regards to: ICU length of stay (LOS), ICU mortality, hospital LOS, and hospital mortality and to assess the acceptability of small phlebotomy tubes in adult ICU and IMU patients.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the medical ICU or IMU.
* Hemoglobin less than 10 g/dL.

Exclusion Criteria:

* Clinical bleeding. Defined as any bleeding needing an intervention. An intervention could be an increase in the frequency of hemoglobin monitoring, a transfusion, a procedure, or a consultation intended to prevent or treat bleeding.
* Hemolytic disorder (e.g. sickle cell disease, hereditary spherocytosis, autoimmune hemolytic anemia).
* Bone marrow disorder (e.g. aplastic anemia, leukemia, marrow infiltration disorder, chemotherapy within the last 8 weeks).
* Jehovah's Witnesses.
* Patient is comfort care measures only.
* Refractory shock: Mean arterial blood pressure below 65 mmHg despite maximal doses of 3 vasopressors. Maximal dose of vasopressors are as follows: Norepinephrine 70 mcg/min; vasopressin 0.03 units/min; epinephrine 35 mcg/min; dopamine 20 mcg/kg/min; phenylephrine 350 mcg/min.
* Severe acidosis: pH below 7 in more than one arterial blood gas in the past 24 hours, in the absence of diabetic ketoacidosis.
* Surgical admission diagnosis.
* Pregnancy.
* Current prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 688 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants that receive a red blood cell (RBC) transfusion during hospitalization | up to 30 days after randomization

SECONDARY OUTCOMES:
Number of RBC units transfused during hospitalization | up to 30 days after randomization
Length of stay in ICU | completion of study (up to 90 days from enrollment)
Number of participants that died while in ICU | completion of study (up to 90 days from enrollment)
Length of stay in hospital | completion of study (up to 90 days from enrollment)
Number of participants that died while in hospital | completion of study (up to 90 days from enrollment)
Acceptability of small tubes as assessed by determining the number of patients that switch from small tubes to standard tubes | up to 30 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Javier Barreda Garcia, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No